CLINICAL TRIAL: NCT02602782
Title: Physiologic Signals and Signatures With the Accuryn™ Monitoring System in Intensive Care Patients
Acronym: PRESCIENT
Status: Completed | Type: Observational
Sponsor: Potrero Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD-06-1346
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Critical Care, Intensive Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

SUMMARY:
The purpose of the study is to collect physiologic data streams with the Accuryn Monitoring System and validate the accuracy of these measurements against existing gold standards, and to track and analyze changes in these physiologic data streams to identify clinical signatures that may enable earlier diagnosis and intervention of critical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the hospital with trauma (including burn)
* Anticipated ICU stay of at least 72 hours
* Anticipated transfusion of ≥1 unit blood products (pRBC's, platelets, and/or plasma) within the first 24 hours of hospitalization, and/or a current diagnosis of sepsis/septic shock, and/or ICU admission primarily for burn
* Anticipated requirement for a urinary bladder catheter for ≥ 72 hours

Exclusion Criteria:

* Inability to receive a 16F urinary bladder catheter
* Significant bladder or urethral injury
* In the opinion of the investigator the patient is unsuitable for the study for any other legitimate reason including incarceration, pre-existing medical or psychiatric condition, or interfering medications
* Known previous or concurrent enrollment in a clinical trial that, in the opinion of the investigator, might interfere with the objectives of this clinical trial
* Pregnancy known at the time of presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Significantly injured trauma ICU patients receiving a Foley catheter and transfusion
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Comparison of physiologic signals as measured by the Accuryn Monitoring System compared to existing gold standard measurements. | During the ICU stay (approximately 2-4 weeks)